CLINICAL TRIAL: NCT01239992
Title: Effect of Niacin/Laropiprant on Postprandial Lipoprotein and Glucose Metabolism in Patients With Severe Dyslipoproteinemia
Brief Title: Effect of Niacin/Laropiprant on Postprandial Lipoprotein Metabolism in Patients With Dyslipoproteinemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: negative endpoint study resulting in withdrawal of study drug
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Klaus Parhofer, Professor of Medicine, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KP-Niacin-2010; 2010-019954-42 (EudraCT Number)
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-03

CONDITIONS: Hyperlipoproteinemia; Metabolic Syndrome
MeSH Terms: conditions — Hyperlipoproteinemias; Metabolic Syndrome | interventions — Niacin; MK-0524

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Niacin/ Laropiprant (Experimental)
  Interventions: Drug: Niacin/ Laropiprant

INTERVENTIONS:
Drug: Niacin/ Laropiprant — 1000/ 20 mg first 4 weeks, 2000/40 mg next 8 weeks; daily
  Other Names: Tredaptive; EU/1/08/459/001

SUMMARY:
The study is designed to evaluate the effect of Niacin/Laropiprant on postprandial lipoprotein metabolism, postprandial glucose metabolism, postprandial monocyte function, and postprandial biomarkers of endothelial dysfunction and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects or postmenopausal female subjects aged between 19-70 years
* High risk patients (PROCAM risk ≥20%) on a stable statin-therapy, but at least simvastatin 20 mg/d
* HDL-cholesterol ≤50 mg/dl and /or triglycerides 150-400 mg/dl and/or LDL-cholesterol 70 - 150 mg/dl
* Lipoprotein (a) < 30 mg/dl
* Patients may have normal glucose metabolism (normal HOMA), be insulin resistant (abnormal HOMA), have impaired fasting glucose or impaired glucose tolerance but not diabetes mellitus.
* Without niacin therapy for at least 6 months
* Dosage of any concomitant medication has been stable for at least 3 weeks
* If female, postmenopausal (absence of menstruation for at least 12 months or absence of menstruation > 6 months with FSH > 40 ng/ml respectively oestrogen < 20 pg/ml)

Exclusion Criteria:

* Subjects with additional causes for hyperlipoproteinemia
* Diabetes mellitus or antidiabetic medication
* Subject has history of cardiovascular ischemia in previous 3 months or acute myocardial infarction or unstable angina
* History of psychiatric disorder or cognitive impairment that would interfere with participation in the study
* History of alcoholism
* Contraindication against niacin and/or laropiprant
* Subject has participated in an investigational study within 30 days prior to study initiation
* Fasting triglycerides >400 mg/dl
* Life-threatening disease (e.g. cancer)
* Renal insufficiency (GFR ≤ 30 ml/min )
* Major hepatic impairment
* Known allergic reaction/intolerance against niacin and/or laropiprant
* Active peptic ulcer disease

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Parhofer, MD, Prof., Principal Investigator — Medizinische Klinik II, Klinikum der Universitaet Muenchen, Grosshadern
Locations (1):
- Medizinische Klinik II, Klinikum der Universitaet Muenchen, Grosshadern, Munich, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Niacin/ Laropiprant
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Niacin/ Laropiprant
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 12

OUTCOME MEASURES:

1. Primary Outcome: Incremental Area Under the Plasma Triglyceride Curve Over 8 Hours Following a Standardized Oral Fat Tolerance Test
Description: Percent change of incremental AUC at 12 weeks compared to baseline.
Time Frame: baseline and 12 weeks after treatment
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Niacin/ Laropiprant
Number analyzed (Participants) | 10
percentage change | -28 (5)

2. Secondary Outcome: HDL Cholesterol
Description: Percent change of HDL-cholesterol at 12 weeks compared to baseline.
Time Frame: baseline and 12 weeks after treatment
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Niacin/ Laropiprant
Number analyzed (Participants) | 10
percentage change | 17 (6)

3. Secondary Outcome: Fasting Triglycerides
Description: Percent change of fasting triglycerides at 12 weeks compared to baseline
Time Frame: baseline and 12 weeks after treatment
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Niacin/ Laropiprant
Number analyzed (Participants) | 10
percentage change | -26 (15)

4. Other Pre Specified Outcome: LDL-cholesterol
Description: Percent change of LDL-cholesterol at 12 weeks compared to baseline
Time Frame: baseline and 12 weeks after treatment
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Niacin/ Laropiprant
Number analyzed (Participants) | 10
percentage change | -20 (8)

ADVERSE EVENTS:
Arm/Group | Niacin/ Laropiprant
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes